CLINICAL TRIAL: NCT06229951
Title: Efficacy of Hydrolyzed Collagen and Undenatured Collagen Type II in Alleviating Pain in Patients With Knee Osteoarthritis
Brief Title: Hydrolyzed Collagen and Undenatured Collagen Type II in OA Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Varah Yuenyongviwat, Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66-304-11-1
Record Dates: First submitted 2024-01-16; First posted 2024-01-29 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; Collagen supplement
MeSH Terms: conditions — Osteoarthritis | interventions — Collagen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen supplement group (Experimental): Patients who have taken 480 mg of hydrolyzed collagen and 20 mg of undenatured type II collagen (in one tablet) 2 tabs a day
  Interventions: Dietary Supplement: Collagen
- Control group (Placebo Comparator): Control patients will take placebo 2 tabs a day
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Collagen — Patients who have taken 480 mg of hydrolyzed collagen and 20 mg of undenatured type II collagen (in one tablet) 2 tabs a day
  Arms: Collagen supplement group
Other: Placebo — Control patients will take placebo 2 tabs a day.
  Arms: Control group

SUMMARY:
Randomized controlled trial

Targeted patients who come to receive treatment for osteoarthritis that meets the research indications will be assigned to a random group by the box of 4 randomization method, with a sequence that is randomly generated by a computer. The groups are divided into two groups:

Group 1: Patients who have taken 480 mg of hydrolyzed collagen and 20 mg of undenatured type II collagen

Group 2: Control patients will take placebo

Primary outcome : Pain level

ELIGIBILITY:
Inclusion Criteria:

* Age: 50-80 years old
* Medial compartment knee osteoarthritis
* Kellgren and Lawrence classification stage 2 -3
* Able to walk without walking aid

Exclusion Criteria:

* History of knee surgery on the study side
* History of intra-articular steroid injection within 6 months prior to study entry
* Systemic arthritis conditions
* Degenerative neurological and muscular conditions in the lower extremities
* Chronic kidney disease with CrCl < 30 ml/min (glomerular filtration rate <60 mL/min/1.73 m2)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Pain (VNRS) | 12 weeks
  Pain level (verbal numerical rating scale :VNRS) - 0 is no pain and 10 is the worst pain

SECONDARY OUTCOMES:
Knee and Osteoarthritis Outcome Score (KOOS) | 12 weeks
  Knee and Osteoarthritis Outcome Score (KOOS) - 100 indicates the best possible results and 0 the worst outcome
Rescue medication | 12 weeks
  Amount of pain medication intake
Patient satisfaction | 12 weeks
  Patient satisfaction (verbal numerical rating scale :VNRS) - (0-10; 0=worst and 10=best)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: Data will become available and for 1 year after publication.
Access Criteria: Open Science Framework (OSF)
URL: https://osf.io

REFERENCES:
- [Derived] Yuenyongviwat V, Anusitviwat C, Tuntarattanapong P, Hongnaparak T, Iamthanaporn K. Efficacy of combined undenatured type II collagen and hydrolysed collagen supplementation in knee osteoarthritis: a randomised controlled trial. Sci Rep. 2025 Sep 2;15(1):32313. doi: 10.1038/s41598-025-17505-0. PMID 40897777